CLINICAL TRIAL: NCT01585025
Title: Obeticholic Acid Treatment in Patients With Bile Acid Diarrhoea: an Open-label, Pilot Study of Mechanisms, Safety and Symptom Response.
Brief Title: Obeticholic Acid in Bile Acid Diarrhoea
Acronym: OBADIAH1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRO1909; 2011-003777-28 (EudraCT Number)
Record Dates: First submitted 2012-04-23; First posted 2012-04-25 (Estimated); Results first posted 2019-09-13 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Primary Bile Acid Malabsorption; Secondary Bile Acid Malabsorption; Chronic Diarrhoea
Keywords: Primary bile acid malabsorption; Secondary bile acid malabsorption; Chronic diarrhoea; Obeticholic acid; SeHCAT; FXR; FGF19
MeSH Terms: conditions — Bile Acid Malabsorption, Primary | interventions — obeticholic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Primary BAD (Experimental): Defined as SeHCAT <10% without other causes such as Crohn's disease and/or ileal resection
  Interventions: Drug: Obeticholic acid
- Secondary BAD (Experimental): With Crohn's disease or ileal resection
  Interventions: Drug: Obeticholic acid
- Idiopathic Diarrhoea Controls (Experimental): Chronic diarrhoea with SeHCAT >15% and no Crohn's or ileal resection
  Interventions: Drug: Obeticholic acid

INTERVENTIONS:
Drug: Obeticholic acid — Day -14 to Day 0 subjects will stop their usual diarrhoeal medication. Day 1 to Day 15 Obeticholic acid 25mg tablet will be administered to subjects once daily in the morning. Day 16 to day 28 normal diarrhoeal medication may be re-commenced.
  Other Names: INT-747; 6 ethyl chenodeoxycholic acid

SUMMARY:
The investigators propose to develop studies of obeticholic acid (OCA) in patients with bile acid diarrhoea. OCA is a semisynthetic bile acid, also known as 6αethylchenodeoxycholic acid or INT747,and is a potent farnesoid X receptor (FXR) agonist. Preliminary data suggests that patients with bile acid diarrhoea have impaired production of the ileal hormone Fibroblast Growth Factor 19 (FGF19). FGF19 is stimulated by FXR agonists, and regulates bile acid synthesis. This study is a pilot, proof-of-concept, open-label study to investigate whether OCA can stimulate FGF19 in bile acid diarrhoea patients to provide a safe and effective treatment.

DETAILED DESCRIPTION:
Bile acid diarrhoea (BAD) is an under-recognised but common condition of chronic watery diarrhoea. BAD may be secondary to ileal disease affecting the reabsorption and the enterohepatic circulation of bile acids (bile acid malabsorption) or can be an idiopathic, primary BAD (PBAD). In work published in 2009, we described a new mechanism to explain this syndrome of primary BAD.

Blood levels of the hormone fibroblast growth factor 19 (FGF19) are reduced in primary and secondary BAD, producing impaired feedback inhibition of bile acid synthesis, leading to excess faecal bile acids, which then produce diarrhoea by stimulating colonic secretion. FGF19 is synthesised in the ileum and we have shown transcription is markedly induced by farnesoid X receptor(FXR) agonists such as chenodeoxycholic acid, an abundant natural bile acid. More potent FXR agonists are logical diagnostic and therapeutic agents for this condition, and obeticholic acid (OCA), which is 100x more potent than chenodeoxycholic acid, has recently been developed. It has been used in phase II studies in primary biliary cirrhosis and in non-alcoholic steatohepatitis where a relatively common side-effect was constipation.

We aim to investigate the effects of OCA in patients with primary and secondary BAD to determine whether FGF19 is able to be stimulated in these conditions. We will compare these responses to those in control patients with chronic diarrhoea but without evidence of BAD. It is possible in BAD that the defect in FGF19 levels is due to an inability to respond to FXR stimulation (particularly likely in secondary BAD after ileal resection). Patients with primary BAD may be able to respond and benefit from an increase in FGF19 levels.

This study aims to obtain pilot data on the effects of OCA on FGF19, other markers of bile acid metabolism and patient symptoms including diarrhoea. These are early phase II, proof of concept studies.

ELIGIBILITY:
Inclusion Criteria Patients aged 18 - 80 who present at routine Gastrointestinal Outpatient Clinics at Hammersmith and Charing Cross Hospitals with chronic diarrhoea, defined as an average stool frequency of at least three per day, of Bristol Stool Type 6 or 7, for at least 3 months. Previous routine SeHCAT testing to establish the presence or absence of bile acid diarrhoea (BAD) unless there is evidence of TI disease/ resection. BAD will be defined as SeHCAT 7-day retention of less than 15% or diarrhoea in presence of TI disease/ resection. Study subjects will be grouped as having secondary BAD, due to ileal resection or Crohn's disease, or primary BAD, with no obvious cause. The third, control group having chronic diarrhoea but with normal SeHCAT retention (greater than 15%).

Female patients must be postmenopausal, surgically sterile, or if premenopausal, be prepared to use ≥ 1 effective (≤ 1% failure rate) method of contraception during the trial and for 15 days after the last dose of OCA. Male subjects with female partners of childbearing potential must use ≥ 1 effective method of contraception. Effective methods of contraception are considered to be: 1. Established use of oral, injected or implanted hormonal methods of contraception. 2. Placement of an intrauterine device (IUD) or intrauterine system (IUS). 3. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository. 4. Male sterilisation (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate). 5. True abstinence: When this is in line with the preferred and usual lifestyle of the subject.

Exclusion Criteria

* Patients with other diagnoses leading to diarrhoea, including colorectal neoplasia, ulcerative colitis, coeliac disease, chronic pancreatitis, drug-induced diarrhoea or active infection.
* Patients who have not been investigated by standard clinical assessments to exclude these disorders.
* Treatment with bile acid sequestrants (colestyramine, colestipol, colesevelam) for 2 weeks before the first dose of OCA. Loperamide use will be allowed up to 16mg/d in divided doses.
* Previous biliary surgery, excluding cholecystectomy.
* Abnormal bilirubin, alanine aminotransferase (ALT), aspartate aminotransferase (AST) or alkaline phosphatase on more than 1 occasion.
* Chronic liver disease
* Chronic kidney disease
* Active, serious medical disease with likely life expectancy less than 5 years
* Active substance abuse including inhaled or injection drugs in the year prior to screening
* Allergy to obeticholic acid.
* Pregnancy, planned pregnancy, potential for pregnancy and unwillingness to use effective birth control during the trial, breast feeding. Pregnancy will be assessed with urinary β-hCG pregnancy test.
* Participation in an investigational new drug trial in the 30 days before randomisation
* Any other condition which, in the opinion of the investigator, would impede compliance or hinder completion of the study
* Failure to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-04; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julian RF Walters, MBBS MA FRCP, Principal Investigator — Imperial College London
Locations (2):
- United Kingdom (2):
  - Hammersmith Hospital, Imperial College Healthcare NHS Trust, London
  - Hammersmith Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wedlake L, A'Hern R, Russell D, Thomas K, Walters JR, Andreyev HJ. Systematic review: the prevalence of idiopathic bile acid malabsorption as diagnosed by SeHCAT scanning in patients with diarrhoea-predominant irritable bowel syndrome. Aliment Pharmacol Ther. 2009 Oct;30(7):707-17. doi: 10.1111/j.1365-2036.2009.04081.x. Epub 2009 Jun 30. PMID 19570102
- [Background] Hofmann AF. The syndrome of ileal disease and the broken enterohepatic circulation: cholerheic enteropathy. Gastroenterology. 1967 Apr;52(4):752-7. No abstract available. PMID 5337211
- [Background] Walters JR, Tasleem AM, Omer OS, Brydon WG, Dew T, le Roux CW. A new mechanism for bile acid diarrhea: defective feedback inhibition of bile acid biosynthesis. Clin Gastroenterol Hepatol. 2009 Nov;7(11):1189-94. doi: 10.1016/j.cgh.2009.04.024. Epub 2009 May 6. PMID 19426836
- [Background] Hofmann AF, Mangelsdorf DJ, Kliewer SA. Chronic diarrhea due to excessive bile acid synthesis and not defective ileal transport: a new syndrome of defective fibroblast growth factor 19 release. Clin Gastroenterol Hepatol. 2009 Nov;7(11):1151-4. doi: 10.1016/j.cgh.2009.07.026. Epub 2009 Aug 7. No abstract available. PMID 19665580
- [Background] Oelkers P, Kirby LC, Heubi JE, Dawson PA. Primary bile acid malabsorption caused by mutations in the ileal sodium-dependent bile acid transporter gene (SLC10A2). J Clin Invest. 1997 Apr 15;99(8):1880-7. doi: 10.1172/JCI119355. PMID 9109432
- [Background] Montagnani M, Love MW, Rossel P, Dawson PA, Qvist P. Absence of dysfunctional ileal sodium-bile acid cotransporter gene mutations in patients with adult-onset idiopathic bile acid malabsorption. Scand J Gastroenterol. 2001 Oct;36(10):1077-80. doi: 10.1080/003655201750422693. PMID 11589382
- [Background] Makishima M, Okamoto AY, Repa JJ, Tu H, Learned RM, Luk A, Hull MV, Lustig KD, Mangelsdorf DJ, Shan B. Identification of a nuclear receptor for bile acids. Science. 1999 May 21;284(5418):1362-5. doi: 10.1126/science.284.5418.1362. PMID 10334992
- [Background] Inagaki T, Choi M, Moschetta A, Peng L, Cummins CL, McDonald JG, Luo G, Jones SA, Goodwin B, Richardson JA, Gerard RD, Repa JJ, Mangelsdorf DJ, Kliewer SA. Fibroblast growth factor 15 functions as an enterohepatic signal to regulate bile acid homeostasis. Cell Metab. 2005 Oct;2(4):217-25. doi: 10.1016/j.cmet.2005.09.001. PMID 16213224
- [Background] Lundasen T, Galman C, Angelin B, Rudling M. Circulating intestinal fibroblast growth factor 19 has a pronounced diurnal variation and modulates hepatic bile acid synthesis in man. J Intern Med. 2006 Dec;260(6):530-6. doi: 10.1111/j.1365-2796.2006.01731.x. PMID 17116003
- [Background] Brydon WG, Nyhlin H, Eastwood MA, Merrick MV. Serum 7 alpha-hydroxy-4-cholesten-3-one and selenohomocholyltaurine (SeHCAT) whole body retention in the assessment of bile acid induced diarrhoea. Eur J Gastroenterol Hepatol. 1996 Feb;8(2):117-23. doi: 10.1097/00042737-199602000-00005. PMID 8723414
- [Background] Johnston I, Nolan J, Pattni SS, Walters JR. New insights into bile acid malabsorption. Curr Gastroenterol Rep. 2011 Oct;13(5):418-25. doi: 10.1007/s11894-011-0219-3. PMID 21805078
- [Derived] Walters JR, Johnston IM, Nolan JD, Vassie C, Pruzanski ME, Shapiro DA. The response of patients with bile acid diarrhoea to the farnesoid X receptor agonist obeticholic acid. Aliment Pharmacol Ther. 2015 Jan;41(1):54-64. doi: 10.1111/apt.12999. Epub 2014 Oct 20. PMID 25329562

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Primary BAD | Secondary BAD | Idiopathic Diarrhoea Controls
Started | 10 | 13 | 12
Completed | 10 | 10 | 8
Not Completed | 0 | 3 | 4
Not completed — Withdrawal by Subject | 0 | 3 | 4

BASELINE CHARACTERISTICS:
Population: Received any dose of medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Primary BAD | Secondary BAD | Idiopathic Diarrhoea Controls | Total
Number analyzed (Participants) | 10 | 10 | 8 | 28
Age, Continuous [Median (Full Range); unit: years] | 47 [24 to 74] | 45 [27 to 71] | 39 [25 to 68] | 41 [24 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 3 | 17
  Male | 3 | 3 | 5 | 11
Region of Enrollment [Number; unit: participants]
  United Kingdom | 10 | 10 | 8 | 28

OUTCOME MEASURES:

1. Primary Outcome: Changes in Fasting FGF19
Description: The primary outcome measure is the change over 2 weeks in fasting serum fibroblast growth factor (FGF19) in 3 groups of patients: primary bile acid diarrhoea, secondary bile acid diarrhoea, and a control population of patients with chronic diarrhoea but with normal bile acid retention.
Time Frame: Day 0, Day 15
Measure: Median (Inter-Quartile Range); unit: percentage increase of baseline
Arm/Group | Primary BAD | Secondary BAD | Idiopathic Diarrhoea Controls
Number analyzed (Participants) | 10 | 10 | 8
percentage increase of baseline | 71 [9 to 102] | 25 [-6 to 140] | 130 [-14 to 304]
Statistical Analysis 1: Comparison: Primary BAD; Paired comparison of fasting FGF19 at baseline on day 0 and on day 14 of OCA treatment; Test type: Superiority; p = 0.007, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Secondary BAD; Paired comparison of fasting FGF19 at baseline on day 0 and on day 14 of OCA treatment; Test type: Superiority; p = 0.11, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Idiopathic Diarrhoea Controls; Paired comparison of fasting FGF19 at baseline on day 0 and on day 14 of OCA treatment; Test type: Superiority; p = 0.12, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Changes in Non-fasting Response of FGF19 to OCA
Description: Change in dynamic response of FGF19 in 6 hours following OCA administration; at start and end of 15 day OCA test period.
Time Frame: Day 0, Day 15
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | Primary BAD | Secondary BAD | Idiopathic Diarrhoea Controls
Number analyzed (Participants) | 10 | 10 | 8
percentage change | 11.6 [-23.6 to 57.8] | 14.6 [-22.7 to 49.0] | 32.4 [15.1 to 38.4]
Statistical Analysis 1: Comparison: Primary BAD; Change in FGF19 AUC; Test type: Superiority; p = 0.72, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Secondary BAD; Change in FGF19 AUC; Test type: Superiority; p = 0.51, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Idiopathic Diarrhoea Controls; Change in FGF19 AUC; Test type: Superiority; p = 0.13, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Changes in Fasting 7α-hydroxy-4-cholesten-3-one
Description: Change in fasting 7α-hydroxy-4-cholesten-3-one before and after 15 day administration of OCA.
Time Frame: Day 0, Day 15
Population: Missing data in Primary BAD
Measure: Median (Inter-Quartile Range); unit: microgram/L
Arm/Group | Primary BAD | Secondary BAD | Idiopathic Diarrhoea Controls
Number analyzed (Participants) | 8 | 10 | 8
microgram/L | -11.5 [-30.0 to -3.5] | -27.5 [-56.3 to 0] | -6.5 [-11.5 to -1.5]
Statistical Analysis 1: Comparison: Primary BAD; Change in fasting C4; Test type: Superiority; p = 0.03, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Secondary BAD; Change in fasting C4; Test type: Superiority; p = 0.11, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Idiopathic Diarrhoea Controls; Change in fasting C4; Test type: Superiority; p = 0.02, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Changes in Serum Total Bile Acids.
Description: Dynamic changes of total bile acids over 6 hour period following OCA administration before and after 15 day OCA period.
Time Frame: Day 0, Day 15
Measure: Median (Inter-Quartile Range); unit: micromol/L
Arm/Group | Primary BAD | Secondary BAD | Idiopathic Diarrhoea Controls
Number analyzed (Participants) | 10 | 10 | 8
micromol/L | -18.1 [-33.0 to -5.50] | -2.0 [-17.5 to 0.08] | -15.5 [-17.9 to -14.0]
Statistical Analysis 1: Comparison: Primary BAD; Change in bile acid 6h AUC; Test type: Superiority; p = 0.02, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Secondary BAD; Change in bile acid 6h AUC; Test type: Superiority; p = 0.04, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Idiopathic Diarrhoea Controls; Change in bile acid 6h AUC; Test type: Superiority; p = 0.02, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Changes in Stool Frequency
Description: Change in total number of stool episodes reported per week between week 2 (baseline) and week 4 (week 2 of treatment)
Time Frame: Week 2, Week 4
Population: Missing data in Idiopathic diarrhoea controls
Measure: Median (Inter-Quartile Range); unit: stools per week
Arm/Group | Primary BAD | Secondary BAD | Idiopathic Diarrhoea Controls
Number analyzed (Participants) | 10 | 10 | 7
stools per week | -4.5 [-9.3 to -1.5] | -2.5 [-15.8 to 1.8] | 3.0 [-3.0 to 7.0]
Statistical Analysis 1: Comparison: Primary BAD; Comparison of change in number of stools per week; Test type: Superiority; p = 0.03, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Secondary BAD; Comparison of change in number of stools per week; Test type: Superiority; p = 0.17, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Idiopathic Diarrhoea Controls; Comparison of change in number of stools per week; Test type: Superiority; p = 0.31, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Changes in Mean Stool Form
Description: Change in mean stool form reported per week between week 2 (baseline) and week 4 (week 2 of treatment) using the Bristol Stool Form Scale (range of scores 1 to 7). High scores are a worse outcome (7=liquid stools).
Time Frame: Week 2, Week 4
Population: Missing data in Idiopathic diarrhoea controls
Measure: Median (Inter-Quartile Range); unit: Score on Bristol scale
Arm/Group | Primary BAD | Secondary BAD | Idiopathic Diarrhoea Controls
Number analyzed (Participants) | 10 | 10 | 7
Score on Bristol scale | -0.71 [-1.54 to 0.10] | -0.38 [-0.91 to -0.18] | -0.46 [-0.91 to 0.86]
Statistical Analysis 1: Comparison: Primary BAD; Change in median stool form; Test type: Superiority; p = 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Secondary BAD; Change in median stool form; Test type: Superiority; p = 0.04, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Idiopathic Diarrhoea Controls; Change in median stool form; Test type: Superiority; p = 0.74, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Change in Stool Index
Description: Change in index calculated on a weekly basis, between week 2 (baseline) and week 4 (week 2 of treatment).
  Index calculated as ([weekly stool frequency x mean Bristol Stool Form Scale score] = Loperamide use [weekly mg x 3]).
  Individual scores ranged from 25 to 1095, with higher scores being worst.
Time Frame: Week 2, Week 4
Population: Missing data in Idiopathic diarrhoea controls
Measure: Median (Inter-Quartile Range); unit: index score
Arm/Group | Primary BAD | Secondary BAD | Idiopathic Diarrhoea Controls
Number analyzed (Participants) | 10 | 10 | 7
index score | -37.5 [-52.3 to -22.8] | -32.5 [-158.6 to -13.4] | -5.5 [-30.0 to 20.0]
Statistical Analysis 1: Comparison: Primary BAD; Paired difference in weekly index score; Test type: Superiority; p = 0.005, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Secondary BAD; Paired difference in weekly index score; Test type: Superiority; p = 0.03, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Idiopathic Diarrhoea Controls; Paired difference in weekly index score; Test type: Superiority; p = 0.61, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Data were collected over the 6 weeks of the trial
Arm/Group | Primary BAD | Secondary BAD | Idiopathic Diarrhoea Controls
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/8
Other Adverse Events (participants affected / at risk) | 0/10 | 3/10 | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary BAD (N=10) | Secondary BAD (N=10) | Idiopathic Diarrhoea Controls (N=8)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Constipation/abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Recruitment in the idiopathic chronic diarrhoea control group did not reach the prespecified number of 10 due to dropouts. Of the 8 subjects recruited, one failed to return diaries that could be analysed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes